CLINICAL TRIAL: NCT00192062
Title: A Phase II Trial of Gemcitabine (Gemzar) Combined With Vinorelbine as First Line Chemotherapy for Metastatic Breast Cancer
Brief Title: A Trial of Gemcitabine Combined With Vinorelbine as First Line Chemotherapy for Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7775; B9E-EY-S372
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-08-31 (Estimated); Status verified 2007-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine; Vinorelbine

INTERVENTIONS:
Drug: gemcitabine
Drug: vinorelbine

SUMMARY:
This is a Phase II study of gemcitabine- Vinorelbine combination in a 3-weekly schedule as first line chemotherapy in patients with metastatic breast cancer. Eighty patients with measurable disease will be enrolled in the study. Gemcitabine will be used at 1000 mg/m2, vinorelbine at 25mg/m2. Every cycle, vinorelbine will be administered before gemcitabine. After the initial dose, modifications of Gemcitabine and vinorelbine doses are allowed based on patient toxicity

Study therapy may continue until:

* There is evidence of progressive disease
* The patient experiences unacceptable toxicity.
* The investigator decides that the patient should be discontinued
* The patient requests discontinuation
* The patient has received 6 cycles of the regimen(if the physician decides to continue after 6 cycles-this will be done after consultation with the sponsor)
* Discontinuation from study therapy is indicated according to the protocol It's the investigator's responsibility to strictly stick to the protocol procedures. It needs to be discussed with Lilly medical designee in advance when any special situation occurs which has not been defined in protocol.

After patients discontinue from study therapy, they proceed to the post-study follow up phase of the study. Assessments to take place during this phase are outlined in the protocol.

ELIGIBILITY:
Inclusion Criteria-

* Histological or cytological diagnosis of breast carcinoma with evidence of unresectable, locally recurrent, or metastatic disease. Lesions should not be amenable to surgery or radiation of curative intent.
* Presence of metastatic or local-regional recurrent disease, according to the American Joint Committee on Cancer (Greenz, et al, 2002).
* Uni-dimensionally measurable lesions with clearly defined margin that are clearly measurable by following methods according to computerized tomography (CT), Chest x-ray or clinical examination, according to RECIST criteria (Therasse, et al, 2002).
* No prior chemotherapy for metastatic or locoregionally recurrent disease. Prior adjuvant or neoadjuvant chemotherapy with Anthracyclines based regimen is mandatory. The time from the last dose of prior adjuvant chemotherapy and study entry must be at least 30 days and patients must have completely recovered from all acute chemotherapy related toxicities (with exception of alopecia).
* Prior radiotherapy must be completed at least 30 days before study entry.
* No concurrent hormonal therapy for MBC. Prior hormonal therapy is allowed, the time from the last dose of prior hormonal therapy for breast cancer to study enrollment must be at least 1 week.

Exclusion Criteria -

* Have received treatment within the last 30 days with an investigational drug for any indication before study entry.
* Concurrent administration of other tumor therapy, including cytotoxic chemotherapy, surgery of cancer, radiotherapy, hormonal therapy and immunotherapy (including Herceptin).
* Active infection that in the opinion of the investigator would compromise the patient's ability to tolerate therapy, unless adequately treated.
* Pregnancy or breast-feeding.
* Serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2004-07; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the response rate of Gemcitabine-vinorelbine when used in a 3-weekly as first line chemotherapy in patients with metastatic breast cancer.

SECONDARY OUTCOMES:
To characterize the quantitative and qualitative toxicity of Gemcitabine-vinorelbine patient population
Relative dose density of Gemcitabine and vinorelbine
Rate of dose modifications (admissions, reductions, delays)
Time to progression
Duration of response
1 year survival

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- Egypt (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Alexandria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Assyout
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Cairo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Giza

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com